CLINICAL TRIAL: NCT03846115
Title: A Technology Solution for Peer-led Seeking Safety
Brief Title: A Mobile App for Peer-led Seeking Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Innovations (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2R44DA041949-02 (NIH); 2R44DA041949-02 (NIH)
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Substance Use Disorders; PTSD; Trauma; Emotional Dysfunction
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-Led Seeking Safety app (Experimental): This app is designed for Peer-Led Seeking Safety and includes enhanced app features.
  Interventions: Behavioral: Peer-Led Seeking Safety app
- Control app (Active Comparator): This is a basic app that controls for time and attention. The basic app serves as the intervention in this trial.
  Interventions: Behavioral: Control app

INTERVENTIONS:
Behavioral: Peer-Led Seeking Safety app — This app offers participants sessions of Seeking Safety plus enhanced app features designed to engage and sustain participants in their recovery work.
  Arms: Peer-Led Seeking Safety app
Behavioral: Control app — This app offers the Seeking Safety content but without the enhanced features
  Arms: Control app

SUMMARY:
Peer support is historically prominent for substance use disorder (SUD), such as the world-wide model of Alcoholics Anonymous and other 12-step groups. Yet for trauma and posttraumatic stress disorder (PTSD) there have been few attempts at peer help. A major challenge of trauma peer groups is that they usually focus on telling the story of members' trauma histories, which can be overly triggering and distressing. Seeking Safety offers an excellent choice for peer-led care. It is an evidence-based and is the most widely adopted model for SUD/PTD. It is present-focused, cognitive-behavioral, and provides psychoeducation and coping skills to help clients attain greater safety in their lives. It has been successfully implemented in peer-led format for many years and has been studied in various trials, including a recent randomized controlled trial (RCT) comparing peer versus professional delivery, with positive results. In Phase 1 we developed a beta version of a mobile app for peer-led Seeking Safety (PLSS). In Phase 2 we will enhance the app features and content and also conduct an RCT in a sample of adults with current SUD/PTSD to compare the Peer Safety app condition to a control app.

DETAILED DESCRIPTION:
Peers are increasingly recognized as an important asset in healthcare. Peer support is historically most prominent for substance use disorder (SUD), such as the world-wide model of Alcoholics Anonymous and other 12-step groups. Yet for trauma and posttraumatic stress disorder (PTSD) there have been few attempts at peer help. A major challenge of trauma peer groups is that they usually focus on telling the story of members' trauma histories, which can be overly triggering and distressing. Seeking Safety offers an excellent choice for peer-led care. It is an evidence-based and is the most widely adopted model for SUD/PTD. It is present-focused, cognitive-behavioral, and provides psychoeducation and coping skills to help clients attain greater safety in their lives-- safety from unsafe behavior toward themselves and others, substance use, and trauma symptoms. It has been successfully implemented in peer-led format for many years and has been studied in various trials, including a recent randomized controlled trial (RCT) comparing peer versus professional delivery, with positive results. In Phase 1 we developed a beta version of a mobile app for peer-led Seeking Safety (PLSS). The Peer Safety (PS) app was based on extensive input from end users and was evaluated in a feasibility study. We found strong positive results in Phase 1 and are now conducting a Phase 2 project to continue this work. In Phase 2 we are enhancing the app features and content and will also conduct an RCT in a sample of adults with current SUD/PTSD to compare the PS app condition to a control app. They will have 12 weeks to use the app and participate in weekly online PLSS, and will be assessed pre, post and at 3-month followup using validated instruments. We will also measure app usage and satisfaction. The primary outcomes are substance use and trauma symptoms. Our public health goal is to leverage technology to create PLSS in an online environment that would support recovery, powered by highly engaging content and delivery. The PS app could address the need for access in remote locations, for anonymous help, and for convenient, low-cost help, delivered by people who share their experiences as peers. Even for those who do attend in-person modalities, the app can provide additional support and unique features. This project proposes a novel technology solution to provide care for an important population-- people with SUD/PTSD.

ELIGIBILITY:
Inclusion Criteria:

* meets DSM-5 criteria for current SUD and current PTSD (the latter either full or subthreshold)
* has a mobile device, either Android or iOS.

Exclusion Criteria:

* current uncontrolled psychotic or bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Change in substance use on the Brief Addiction Monitor | Baseline, end of intervention (12 weeks), 3 months after end of intervention
  Past 30 days substance use and related problems
Change in trauma symptoms | Baseline, end of intervention (12 weeks), 3 months after end of intervention
  Trauma Symptom Checklist 40

SECONDARY OUTCOMES:
Amount of time spent on the app | Baseline, end of intervention (12 weeks)
  App usage data
Change in coping self-efficacy on the Coping Self-Efficacy Scale | Baseline, end of intervention (12 weeks), 3 months after end of intervention
  Higher scores indicate stronger perceived ability to cope with challenges; scaling is 0 ('cannot do at all'), 5 ('moderately certain can do') and 10 ('certain can do'). An overall score is computed by summing all items.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Najavits, PhD, Principal Investigator — Treatment Innovations
Locations (1):
- Treatment Innovations, Newton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No